CLINICAL TRIAL: NCT06514391
Title: Immediate Loading of Four Single Piece Compressive Implants for Bar Retained Mandibular Overdenture: A Study of Peri Implant Soft Tissue Health and Marginal Bone Loss
Brief Title: Immediate Loading of Four Single Piece Compressive Implants for Bar Retained Mandibular Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed shady, Assistant Professor, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A14030123
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Compressive Implants

STUDY DESIGN:
Intervention Model Description: all patients recieved 4 inter-foraminal compressive single piece dental implants in the mandible, then milled bar was digitally constructed and cemented to 4 implants to support mandibular implant overdenture
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- compressive one piece implants with bar attachment (Experimental): All patients received 4 mandibular inter-foraminal single piece compressive implants, bar attachment connecting 4 implants was then cemented and complete mandibular overdenture was attached to bar via peek clips
  Interventions: Procedure: compressive single piece dental implant

INTERVENTIONS:
Procedure: compressive single piece dental implant — 4 inter-foraminal single piece compressive dental implants were placed in the mandible via flapless protocol by the aid of stereolithographic surgical guide

SUMMARY:
this study was done to evaluate clinically and radiographically four single piece inter-foraminal compressive implant connected via digitally designed co-cr milled bar with distal cantilever supporting mandibular overdenture. The evaluation will be done clinically and radiographically as following:

* Marginal bone loss
* Soft tissue changes around the implants

DETAILED DESCRIPTION:
Six patients of age ranging from 40 to 60years (mean 50 years) were selected for this study from the out patients clinic, Prosthodontics department, Faculty of Dentistry, Mansoura University.

I) Preparation of the patient for implant placement:

1. A cone beam C.T was done for each patient to determine the bone height and the adequate sites for the placement of four interforaminal implants.
2. Mandibular denture was constructed to aid in designing of surgical stent to guide in implant placement.

II) Surgical phase :

1. Surgical stent was used to guide in implant placement. All implants were placed according to the flapless protocol under local anesthesia.
2. All patients received four dental implants located anterior to the mental foramen in canine and premolar position.

III) Prosthetic phase:

1. The necks of the placed implants were bent up to 15 degree to ensure parallelism.
2. Intraoral final impression was done by intraoral scanner to be used for digital designing of the milled bar and the final prosthesis.
3. bar design was milled in PMMA resin material and tried over implants, then resin bar try-in was invested and casted in co-cr alloy.
4. Final bar was inserted intra-orally after finishing and polishing
5. The four implant bar assembly was then loaded by the prefabricated acrylic denture according to Browaeys H et al , 2014. Access holes were made above the abutment to be finally relined in the patient mouth at the correct vertical dimension of occlusion to allow for immediate loading protocol.
6. The occlusion was adjusted and the patients were instructed to go on soft diet for the first 48 hours until final impressions and delivery of milled bar overdenture were done.

IV) Evaluation:

Probing depth was measured for each implant using plastic probe and radiographic evaluation of the peri-implant marginal bone loss by using cone beam CT started for the patients from the delivery of final prosthesis (T0) and continue for 6 months (T6) and 12 month (T12) from insertion.

ELIGIBILITY:
Inclusion Criteria:

* They were healthy, free from any systemic diseases relating to the bone resorption such as uncontrolled diabetics or osteoprosis .This was achieved through medical history and clinical examination by physician.
* They have completely edentulous maxilla opposed by completely edentulous mandible
* All patients have sufficient inter-arch space for overdenture and milled bar construction not less than 12mm
* All patients are of Angel's class I maxillo-mandibular relationship.
* All patients must have mandibular bone height interforaminally not less than 8-10 mm as verified by cone beam C.T.

Exclusion Criteria:

* Patients with systemic issues such as recent myocardial infarction, hepatic patients, bleeding disorders, autoimmune diseases, hyperparathyroidism
* Uncontrolled diabetes mellitus
* Severe osteoporosis
* Cancer
* Recent organ transplants, long-term corticosteroid use
* Radiotherapy
* Uncooperative patients with psychiatric disorders
* Heavy smokers
* Poor oral hygiene
* Parafunctional habits

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Peri-implant marginal bone loss | at time of insertion of prosthesis T(0), 6 months after insertion T(6), 12 months after insertion T(12)
  Peri-implant marginal bone loss was evaluated for each implant by the aid of cone beam CT scan

SECONDARY OUTCOMES:
Peri-implant soft tissue health | at time of insertion of prosthesis T(0), 6 months after insertion T(6), 12 months after insertion T(12)
  probing depth was measured for each implant by the aid of plastic probe

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shady, MD, Principal Investigator — Mansoura University Faculty of Dentistry, Prosthodontics department
Locations (1):
- Mansoura University, Faculty of dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No